CLINICAL TRIAL: NCT04763720
Title: Implementation of Dyadic Developmental Psychotherapy for Children and Their Families in an Outpatient Setting.
Brief Title: Implementing Dyadic Developmental Psychotherapy (DDP) - Evaluation Research
Status: Enrolling by invitation | Type: Observational
Sponsor: Sykehuset Telemark (Other Government)
Responsible Party: Sponsor
Other Study IDs: 75120X
Record Dates: First submitted 2021-02-02; First posted 2021-02-21 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Psychiatric Problem; Child Neglect; Maltreatment; Child Behavior Problem; DDP
Keywords: Attachment; Dyadic Developmental Psychotherapy; Trauma; Therapy
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dyadic Developmental Psychotherapy: Families being treated with DDP at either of the centres
  Interventions: Behavioral: Dyadic Developmental Psychotherapy

INTERVENTIONS:
Behavioral: Dyadic Developmental Psychotherapy — DDP involves approximately twenty sessions with the family, conducted by a trained DDP therapist. DDP is developed to treat trauma-related and attachment difficulties. DDP is not a manualized treatment but involves using a set of core communication techniques (termed PACE; Playfulness, Acceptance, Curiosity and Empathy).
  Other Names: DDP

SUMMARY:
The objective of this study is to evaluate the implementation and use of Dyadic Developmental Psychotherapy (DDP) in three centra, with particular focus on its potential effects on the quality of the observable caregiver-child interaction. The three centra included are Telemark Hospital Trust, Department for Child- and Adolescent Psychiatric Health, Child Protective Services in Skien and Child Protective Services in Porsgrunn. The implementation of DDP is being led by Telemark Hospital Trust, while therapists from all centra are being trained in DDP as part of the implementation process.

Primarily we aim to identify any changes associated with DDP treatment in the caregiver-child interaction, as measured by the Emotional Availability Scales (EA scales). Our secondary outcome measures assess changes in parental self-efficacy, parental stress, and child emotional and behavioral problems.

The research aims are divided in three research questions:

Q1: What changes are associated with DDP treatment:

Q1.1 the quality of the caregiver-child interaction Q1.2 parental self-efficacy Q1.3 parental stress, Q1.4 child emotional and behavioral problems Based on previous literature, we hypothesize that we will see an increase in the quality of the caregiver-child interaction and parental self-efficacy after completing the DDP treatment, and a decrease in parental stress and child emotional and behavioral problems (Becker-Weidman, A. 2006)

In addition to assessing the effects of DDP we will evaluate the implementation of DDP in the three centra, and inform the implementation by collecting information through interviews with patients and clinicians. We aim to answer:

Q2: How do children and their caregivers experience DDP as a therapeutic intervention? Q3: How do clinicians experience the training process and the use of DDP as a therapeutic intervention?

Based on previous literature, we hypothesize that we will see an increase in the quality of the caregiver-child interaction and parental self-efficacy after completing the DDP treatment, and a decrease in parental stress and child emotional and behavioral problems

DETAILED DESCRIPTION:
Children who have been subject to physical, sexual or emotional abuse or neglect are at risk of developing unhealthy relationships with their caregiver, increasing the likelihood of them developing a wide range of mental health problems later in life. Norway offers few therapeutic programs for treatment of children and adolescents that focus specifically on treating traumatic experiences within attachment relationships. An intervention with this focus is Dyadic Developmental Psychotherapy (DDP),where dyad refers to the unit of a child and its caregiver(s).

The Family-Based Treatment Unit (SFB) within the Division for Child- and Adolescent Mental Health (ABUP) at Telemark Hospital has started implementing DDP with funding from the "BUP Project", resulting in a multi-center implementation plan including local child protective services and the office for children, youth and family affairs. This project seeks to evaluate the implementation of DDP and assess any change in the quality of the caregiver-child interaction, parental efficacy, parental stress and wellbeing, and child emotional and behavioral problems as well as the subjective experience of this implementation among caregivers and clinicians. The results of interviews with clinicians and parents will provide feedback, guide the implementation, and provide essential knowledge about using DDP in a Norwegian setting.

Child protective services (CPS) in the municipalities of Skien and Porsgrunn will be implementing DDP in their respective services and their experiences with the process will also be collected. Mixed method assessment will be used to follow the implementation process.

The present study will contribute new knowledge of how the intervention is experienced by Norwegian children and their families, both in a clinical outpatient setting at Telemark Hospital as well as Skien and Porsgrunn Child Protective Services.

Clinicians' experiences with the implementation and use of DDP is an important dimension for its success.The project will report on what challenges arose during implementation in Norway, and how both families and clinicians experienced the process of learning, using and receiving DDP. By using the information gained directly into the process of this project it can help guide the continued implementation and contribute to its success. If DDP is shown to be a positive and helpful therapeutic methods there are plans for a multi-center randomized controlled trial.

We will investigate the specific context through participant-observations during project meetings, and analyze central documents regarding the implementation and use of DDP.

Through working closely with Child Protective Services we will also be able to explore the experiences of implementation of the treatment in different settings.

Ethical review has been conducted by the Norwegian South East Regional committee for Medical and Health Research (REK) as well as the Norwegian Centre for Research Data (NSD) and the project has been approved. The participants will receive full information, and be asked to give consent both verbally and in writing. They will be assured confidentiality and anonymity. They will be informed of their right to withdraw at any time, and that it will have no impact on their treatment at ABUP. We do not expect this study to cause any harm to participants. The observations are part of routine examination, of short duration and are conducted within the security of a familiar institution

ELIGIBILITY:
Inclusion criteria for child:

1. Symptoms of relational and/or attachment difficulties
2. History of trauma, including neglect or emotional abuse
3. Age 5-18
4. Can understand and make oneself understood in Norwegian

Exclusion criteria for dyad (caregiver and child):

1. Current substance abuse in child or caregiver
2. Current psychosis in child or caregiver
3. Intellectual disability in caregiver Variables that will be tracked but that are not grounds for exclusion are diagnostic variables, including the presence of autism-spectrum disorders, and care-level.

Inclusion criteria for therapists:

1. Trained in DDP
2. Working with DDP in either of the centra

Ages: 5 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Families receiving DDP treatment at any of the centra, that fulfill the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2028-02-29 (Estimated); Study Completion 2028-02-29 (Estimated)

PRIMARY OUTCOMES:
Change in quality of caregiver-child interaction | Time 1 is when the family is referred to DDP treatment, time 2 when treatment is finished, approximately 24 weeks later
  The quality of caregiver-child interaction using the "Emotional Availability Scales". Max total score is 29 and a higher score means better quality interaction.

SECONDARY OUTCOMES:
Change in measured parental self-efficacy | Time 1 is when the family is referred to DDP treatment, time 2 when treatment is finished, approximately 24 weeks later
  Measure of change in parental self-efficacy/competency as measured by the "Parenting Sense of Competence" scale. Max score 96, higher score indicates higher perceived competence.
Change in parental stress | Time 1 is when the family is referred to DDP treatment, time 2 when treatment is finished, approximately 24 weeks later
  Measure of change in parental stress as measured by the "Parental Stress Scale". Max score is 90 and a higher score indicates higher parental stress.
Change in child symptoms of traumatic stress | Time 1 is when the family is referred to DDP treatment, time 2 when treatment is finished, approximately 24 weeks later
  Measure of child's symptoms of traumatic stress as measured by "Child and Adolescent Trauma Screening". Max score is 60, higher score indicates higher levels of traumatic stress.
Change in child emotional and behavioral symptoms | Time 1 is when the family is referred to DDP treatment, time 2 when treatment is finished, approximately 24 weeks later
  General screening of child's symptoms of emotional and behavioral problems, as measured by the "ASEBA" (Achenbach System of Empirically Based Assessment) Child Behavior Checklist. ASEBA uses standardized scores according to age-specific norms, where higher t-scores indicates more/stronger symptoms on each subscale.

OTHER OUTCOMES:
Caregiver's experience of receiving DDP | Approximately 24 weeks after the family has been referred to DDP treatment
  Semi-structured interview exploring the caregiver's experience receiving DDP treatment
Therapists experience of the implementation and use of DDP | Up to every 3rd month after the therapist has been trained in DDP, until the end of the data collection period (31.12.2023)
  Semi-structured focus-group interviews with DDP therapists exploring their experience with the implementation and use of DDP

CONTACTS AND LOCATIONS:
Overall Officials: Idun Røseth, Ph.D, Principal Investigator — Telemark Hospital Trust - University of South-East Norway
Locations (1):
- Telemark Hospital Trust, Skien, Vestfold Og Telemark, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Becker-Weidman A. Treatment for Children with Reactive Attachment Disorder: Dyadic Developmental Psychotherapy. Child Adolesc Ment Health. 2008 Feb;13(1):52. doi: 10.1111/j.1475-3588.2006.00428.x. No abstract available. PMID 32847154